CLINICAL TRIAL: NCT01738750
Title: Laparoscopic Versus Open Appendectomy? Let the Patient Decide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: UU56320
Record Dates: First submitted 2012-11-22; First posted 2012-11-30 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Appendicitis
Keywords: surgical choice; cost of care; decision making; health care; health care cost; pediatric; children; appendicitis; patient satisfaction
MeSH Terms: conditions — Appendicitis; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cost Information Included (Experimental): Group of patients that will receive cost information for both the laparoscopic and open surgical procedures prior to choice of procedure.
  Interventions: Other: Cost Information Included
- No Cost Information Included (No Intervention): Group of patients that will not receive cost information for the laparoscopic and open surgical procedures prior to choice of procedure.

INTERVENTIONS:
Other: Cost Information Included
  Arms: Cost Information Included

SUMMARY:
This protocol examines choice where it pertains to choosing between two standard methods for appendectomy, laparoscopic or open procedures, and the affect that "cost" of the appendectomy has upon choice.

Children admitted with a diagnosis of uncomplicated appendicitis will be consented to participate in a study in which the patient can choose between laparoscopic or open appendectomy procedures. Those that agree to review a consent form will be randomly placed into one of two groups. The two groups consist of one in which the consent form includes "cost information for each operative procedure" in the comparison between the procedures, and the other group receives a consent form that does not include "cost information for each operative procedure". Both groups also view a short, group specific, computerized presentation that describes each procedure.

The hypothesis is that those patients given a choice between two similar surgical procedures and are provided with "cost information" will more often choose the less expensive surgical procedure than those that do not have information related to the cost of the surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* acute appendicitis

Exclusion Criteria:

* age 18 or older
* imaging positive for perforation; ultrasound or CT scan
* pain for greater than 2 days
* children with a body mass index > 95% for age and sex
* surgeon decision for non-equivalent procedure based on patient presentation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Scaife, MD, Principal Investigator — University of Utah
Locations (1):
- Primary Children's Hospital, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Russell KW, Rollins MD, Barnhart DC, Mone MC, Meyers RL, Skarda DE, Soukup ES, Black RE, Molitor MS, Stoddard GJ, Scaife ER. Charge Awareness Affects Treatment Choice: Prospective Randomized Trial in Pediatric Appendectomy. Ann Surg. 2015 Jul;262(1):189-93. doi: 10.1097/SLA.0000000000000885. PMID 25185471

RESULTS

PARTICIPANT FLOW:
Groups:
- Cost Information Included: Group of patients that will receive cost information for both the laparoscopic and open surgical procedures prior to choice of procedure.
  Cost Information Included
Period: Overall Study
Arm/Group | Cost Information Included | No Cost Information Included
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age, Gender
Groups:
- Total: Total of all reporting groups
Arm/Group | Cost Information Included | No Cost Information Included | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (3.3) | 10.6 (3.2) | 10.7 (3.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 51 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 27 | 31 | 58
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Choice Based on Cost
Description: The group given information related to the cost of each surgical procedure will more often choose the less expensive procedure as compared to those not given cost information
Time Frame: Outcome assessed prior to surgical procedure with data presented within 1 year
Measure: Number; unit: percentage of open appendectomy
Groups:
- Cost Information Included; No Cost Information Included: Percentage of Participants who Choose Open Appendectomy or Laparoscopic Appendectomy
Arm/Group | Cost Information Included | No Cost Information Included
Number analyzed (Participants) | 49 | 51
percentage of open appendectomy | 63 | 35

2. Secondary Outcome: Hospital/Operative Dollars
Description: A comparison of the overall hospital admission and operative dollars for acute appendicitis and appendectomy between the two groups
Time Frame: Data will be collected within an expected average of 3 months post-discharge with data presented within 1 year
Measure: Median (Inter-Quartile Range); unit: Dollar
Groups:
- Dollar Information Included: Group of patients that will receive dollars information for both the laparoscopic and open surgical procedures prior to choice of procedure.
  Dollars Information Included
- No Dollar Information Included: Group of patients that will not receive dollar information for the laparoscopic and open surgical procedures prior to choice of procedure.
Arm/Group | Dollar Information Included | No Dollar Information Included
Number analyzed (Participants) | 49 | 51
Dollar | 9,949 [8,601 to 11,338] | 10,477 [9,213 to 11,972]

ADVERSE EVENTS:
Arm/Group | Cost Information Included | No Cost Information Included
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes